CLINICAL TRIAL: NCT05187234
Title: The Effect of Education on Fluid Management, Symptom Control and Quality of Life ın Hemodialysis Patients According to Roy Adaptation Model
Brief Title: The Effect of Education Hemodialysis Patients According to Roy Adaptation Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Özlem Özdemir, PhD, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KırklareliU
Record Dates: First submitted 2021-12-24; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Hemodialysis
Keywords: fluid management,symptom control,life quality
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): Experimental: intervention group The patients were interviewed 3 times, initially at the 1st month and at the 3rd month. All forms were initially administered to patients in the intervention group. Patients were randomly assigned to the intervention group and participated in a one-on-one Roy Adaptation Model-based training program consisting of an initial 30-45 minute session. Hemodialysis Patient Education Manual prepared by the researchers was applied to the patients in the intervention group during the training. All forms were re-administered to the patients in the intervention group in the 1st and 3rd months.
  Interventions: Other: Education
- Control (No Intervention): Education and training manual based on the Roy adaptation model was not given to the patients.

INTERVENTIONS:
Other: Education — Experimental: intervention group Education and training booklet based on the Roy adaptation model was given to the patients. The training was repeated at the first welcome and after the first month.
  Arms: Education

SUMMARY:
The study was conducted in order to evaluate the effect of the training provided to hemodialysis patients according to Roy Adaptation Model on fluid management, symptom control, and quality of life. The study was carried out as a randomized controlled trial with the participation of 107 patients (53 experimental, 54 control) The patients in the experimental group were provided with training based on Roy Adaptation Model, and training booklets were handed out.The control group did not attempt any intervention.

DETAILED DESCRIPTION:
The most difficult domain for hemodialysis patients is fluid-salt restriction. Patients with inadequate fluid compliance/adherence experience many symptoms that negatively affect their life.

The study was carried out as a randomized controlled trial with the participation of 107 patients (53 experimental, 54 control).

The data were collected by using "Patient Information From", "Fluid Control in Hemodialysis Patients Scale" (FCHPS), "Dialysis Symptom Index" (DSI), and "Nottingham Health Profile" (NHP). The forms were filled out by having interviews with the patients in the experimental and control groups in the 0th, 1st, and 3rd months. The patients in the experimental group were provided with training based (face to face individual) on Roy Adaptation Model (0th(onset)and 1st month), and training booklets were handed out. The Training was about 30-45 minutes. control group did not attempt any intervention. Routine maintenance of the control and experimental group and continued. When comparing the experimental and control groups, onset 0th month, 1st month and 3rd month measurements were taken into consideration. All scales were administered to the experimental and control groups at month 0 (onset), 1 and 3 months.

The data were analyzed by using descriptive statistics methods with NCSS (Number Cruncher Statistical System) 2007 software, Student's t-test, Mann-Whitney U Test, Pearson Chi-square test, Fisher-Freeman-Halton Exact test, Repeated Measures test, Bonferroni testi Significance was accepted as p<0,05.

ELIGIBILITY:
Inclusion Criteria:

Patients with end-stage chronic kidney disease older than 18 years undergoing routine hemodialysis treatment for at least 3 months having 3 hemodialysis sessions literate volunteered to participate in the study

Exclusion Criteria:

Patients with acute renal failure previously diagnosed with liver failure and/or malignancy

,patients with New York Heart Society class 3-4 heart failure a history of kidney transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline fluid control | At the end of the 1.st and 3 rd month
  Evaluated by "Fluid Control Scale in Hemodialysis Patients". the scale. The lowest score obtained from the scale was 24 and the highest score was 72, and the higher the score, the greater the compliance of the patients with fluid control.
Change from baseline in symptom severity in patients | At the end of the 1.st and 3 rd month
  Evaluated by 'Dialysis Symptom Index' Using this scoring system, the minimum possible total severity score was 0 if none of the 30 symptoms was present and the maximum potential. Score was 150 if all of the 30 symptoms were reported and rated as "very much bothersome". The minimum value is "0" and the maximum value is "150".
change from baseline quality of life in patients | At the end of the 1.st and 3 rd month
  Evaluated by' Nottingham Health Profile'. It includes 38 items divided into six categories: sleep, physical mobility, energy, pain, emotional reactions, and social isolation. for each of the sections range between 0 ('worst health') and 100 ('best health').

SECONDARY OUTCOMES:
change from baseline ıntradialytic Weight Gain | At the end of the 1.st and 3 rd month
  Interdialytic weight gain was defined as the difference between the predialytic weight and weight at the end of the previous dialysis session

CONTACTS AND LOCATIONS:
Locations (1):
- Kırklareli University, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No